CLINICAL TRIAL: NCT00328042
Title: A Self-Management Intervention for Veterans With Hepatitis C
Brief Title: Hepatitis C Self-Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IAC 05-067
Record Dates: First submitted 2006-05-17; First posted 2006-05-19 (Estimated); Results first posted 2014-09-25 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2014-07

CONDITIONS: Hepatitis C; Chronic Disease
Keywords: Self-care; Quality of Life; Chronic disease
MeSH Terms: conditions — Hepatitis C; Chronic Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-Management Workshop (Experimental)
  Interventions: Behavioral: Self-Management Workshop
- Information Only (Active Comparator)
  Interventions: Behavioral: Information Only

INTERVENTIONS:
Behavioral: Self-Management Workshop — The workshop is a once per week 2.5 hour group that meets for six weeks.
  Arms: Self-Management Workshop
Behavioral: Information Only — This is an individual self-paced at home study program.
  Arms: Information Only

SUMMARY:
The objective of this study is to compare the efficacy of a 6-session hepatitis C self-management workshop to a hepatitis C self-management self-study program. Both interventions are designed to help people with hepatitis C learn to actively self-manage their chronic HCV infection, and ultimately, to improve health outcomes for veterans with HCV who are not receiving Interferon-based treatment. Participants complete a total of four assessments. The fourth assessment, a 12-18 month assessment is an approved addition to the original study design

DETAILED DESCRIPTION:
Background: Chronic hepatitis C (HCV) is a major health concern that disproportionately affects U.S. veterans. Veterans with HCV experience impaired quality of life as a result of HCV infection and other co-morbid disorders; namely substance abuse and mental health problems. Only a small proportion of these patients currently receive and are cured of HCV with Interferon-based treatments. Treatment recommendations for HCV-infected veterans not scheduled for Interferon-based treatment include additional evaluations/procedures and adherence to behavioral/lifestyle guidelines. However, many patients with HCV and commonly occurring co-morbidities have difficulty following these recommendations without additional assistance. HCV self-management programs are one option for helping these patients adhere to treatment recommendations while improving their quality of life. Patient self-management programs augment traditional information-oriented patient education with problem-solving skills and cognitive-behavioral techniques that enable patients to manage chronic illness and their lives as a whole.

Objectives: Our primary objective was to assess the efficacy of a 6-session self-management workshop designed to improve health outcomes for veterans with HCV who are not receiving Interferon-based treatment.

Methods: One hundred- thirty seven Veterans with HCV who receive health care at VA San Diego Healthcare System facilities were randomized to either the HCV Self-Management Workshop (HCV-SMW) or to the Information intervention study arm. The self-management intervention includes six 2.5-hour weekly workshop sessions in addition to the basic information provided to Usual Care. The HCV-SMW was co-led by a health educator and a peer-leader, and has been adapted from an existing self-management program that has been effective for patients with other chronic illnesses. The primary outcome for the study is health-related quality of life. Secondary outcome variables include attendance at recommended health care visits, self-reported health behaviors related to preventing viral transmission, substance use/abuse, and patient-provider communication. Data was collected at baseline, end-of-intervention (6 weeks), at a 12-month and 18-month follow-up visits using self-report questionnaires. In accordance with HIPAA guidelines, VA medical records and other databases were accessed to gather data on health care utilization and mortality. Data was analyzed using repeated-measures analysis of variance, ANCOVA, and linear mixed-model approaches. In addition, an exploratory cost analysis will be conducted when final analyses are conducted.

Status: The study was completed in 2011. Results have been published and citations are provided on this website. An additional manuscript including a cost-effectiveness analysis is in the process of being published.

ELIGIBILITY:
Inclusion Criteria:

* VA patient
* Diagnosis of chronic hepatitis C viral infection

Exclusion Criteria:

* Undergoing treatment with Interferon and/or Ribavirin currently or within 6 months of enrollment
* Inability to confirm HCV diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2007-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik J Groessl, PhD BA BS, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

REFERENCES:
- [Result] Groessl EJ, Weingart KR, Stepnowsky CJ, Gifford AL, Asch SM, Ho SB. The hepatitis C self-management programme: a randomized controlled trial. J Viral Hepat. 2011 May;18(5):358-68. doi: 10.1111/j.1365-2893.2010.01328.x. PMID 20529203
- [Result] Groessl EJ, Weingart KR, Gifford AL, Asch SM, Ho SB. Development of the hepatitis C self-management program. Patient Educ Couns. 2011 May;83(2):252-5. doi: 10.1016/j.pec.2010.06.006. Epub 2010 Jul 17. PMID 20638216
- [Result] Dieperink E, Ho SB, Heit S, Durfee JM, Thuras P, Willenbring ML. Significant reductions in drinking following brief alcohol treatment provided in a hepatitis C clinic. Psychosomatics. 2010 Mar-Apr;51(2):149-56. doi: 10.1176/appi.psy.51.2.149. PMID 20332290
- [Result] Pichetshote N, Groessl E, Yee H, Ho SB. Optimizing the dose and duration of therapy for chronic hepatitis C. Gut Liver. 2009 Mar;3(1):1-13. doi: 10.5009/gnl.2009.3.1.1. Epub 2009 Mar 31. PMID 20479894
- [Result] Groessl EJ, Weingart KR, Kaplan RM, Clark JA, Gifford AL, Ho SB. Living with hepatitis C: qualitative interviews with hepatitis C-infected veterans. J Gen Intern Med. 2008 Dec;23(12):1959-65. doi: 10.1007/s11606-008-0790-y. Epub 2008 Sep 20. PMID 18807097
- [Result] Groessl EJ, Ho SB, Asch SM, Stepnowsky CJ, Laurent D, Gifford AL. The hepatitis C self-management program: sustainability of primary outcomes at 1 year. Health Educ Behav. 2013 Dec;40(6):730-40. doi: 10.1177/1090198113477112. Epub 2013 Feb 27. PMID 23445604
- [Derived] Groessl EJ, Sklar M, Laurent DD, Lorig K, Ganiats TG, Ho SB. Cost-Effectiveness of the Hepatitis C Self-Management Program. Health Educ Behav. 2017 Feb;44(1):113-122. doi: 10.1177/1090198116639239. Epub 2016 Jul 9. PMID 27206463

RESULTS

PARTICIPANT FLOW:
Groups:
- Self-Management Workshop: Self-Management Workshop: In addition to receiving HCV information materials to take home, the in-person 2.5 hour group workshop occurs weekly for six weeks.
- Information Only: Information Only: This group receives a Hepatitis C Information Booklet and an HCV Resource Guide. The materials are designed for individual self-study.
Period: Overall Study
Arm/Group | Self-Management Workshop | Information Only
Started | 69 | 65
Completed | 69 | 63
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Self-Management Workshop: The workshop is a once per week 2.5 hour group that meets for six weeks.
- Arm 2: Self-management self-study: This is an individual self-paced at home study program.
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 69 | 65 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (5.2) | 56.4 (7.2) | 54.6 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 67 | 63 | 130
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 19 | 33
  White | 50 | 42 | 92
  More than one race | 4 | 1 | 5
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 61 | 60 | 121
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 69 | 65 | 134

OUTCOME MEASURES:

1. Primary Outcome: Quality of Well-being Scale - Self-Administered (QWB-SA)
Description: The QWB-SA is a preference-based measure of health-related quality of life. Scores range from 0 to 1.0, with 0 representing death, and 1.0 representing asymptomatic, optimal functioning. Thus, higher scores indicate higher quality of life.
Time Frame: Base Line, 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 69 | 63
units on a scale
  Baseline QWB-SA score | .534 (.153) | .501 (.163)
  12-month QWB-SA score | .600 (.170) | .504 (.152)

2. Secondary Outcome: Hepatitis C Knowledge Questionnaire
Description: The measure consists of 15 questions covering Hepatitis C-specific information related to disease self-management. Each correct response is scored as one point, with total scores range from 0 to 15. Higher scores indicate higher levels of Hepatitis C-specific knowledge. There are no subscales.
Time Frame: Base Line, 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Self-Management Workshop | Information Only
Number analyzed (Participants) | 69 | 63
units on a scale
  Baseline HCV Knowledge | 8.74 (3.12) | 8.60 (2.71)
  6-weeks HCV Knowledge | 12.29 (2.16) | 9.92 (2.75)

ADVERSE EVENTS:
Description: Adverse Events were not monitored for the study as required by the IRB. This was determined because the intervention was considered low risk and consisted of an educational and behavioral change workshop.
Groups:
- Information-Only: Information Only: This group receives a Hepatitis C Information Booklet and an HCV Resource Guide. The materials are designed for individual self-study.
Arm/Group | Self-Management Workshop | Information-Only
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes